CLINICAL TRIAL: NCT02287649
Title: Fc Gamma RIIIA V/F158 Polymorphism and Auto-reactive B and T Cells Subsets in Adult's Immune Thrombocytopenia (ITP) and Correlations With Treatment
Brief Title: Polymorphism and Auto-reactive B and T Cells Subsets in Adult's Immune Thrombocytopenia (ITP)
Acronym: Poly-ITP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P100119
Record Dates: First submitted 2014-11-06; First posted 2014-11-11 (Estimated); Last update posted 2017-10-19 (Actual); Status verified 2017-10

CONDITIONS: Immune Thrombocytopenia
Keywords: Immune thrombocytopenia; Fc gamma RIIIA V/F158 polymorphism; Rituximab; autoreactive B and T cells; ITP
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- patients with rituximab treatment (Other): blood sample intake
  Interventions: Other: blood sample

INTERVENTIONS:
Other: blood sample

SUMMARY:
Aims of the study : 1) To determine whether the presence of the V158 allele of Fc gammaRIIIA gene is associated with a better outcome of Immune Thrombocytopenia (ITP) in adults and especially with a higher response-rate to rituximab. 2) To analyze the impact of therapy and especially rituximab on some B and T cells autoreactive subsets in the peripheral blood.

Patients and Methods :

Inclusion criteria : age ≥ 18 years, primary ITP defined according to the recent consensual criteria (Rodeghiero F et al. Blood 2009), active ITP defined as an ITP with a platelet count < 50 x 109/L requiring treatment, informed consent. Main exclusion criteria : secondary ITP.

Blood samples (serum, plasma, DNA) will be collected in every patient at time of inclusion (pre-treatment) and then sequentially at 3, 6 and 12 months after inclusion in patients treated with rituximab or during the remission phase for other treatments for immunological studies. When a marrow analysis is indicated, some marrow specimens will also be collected and studied and if a patient will have to undergo a splenectomy as a standard of care, some spleen specimens will also be collected. Fc gamma RIIIA V/F158 polymorphism will be assessed by means of an allele-specific PCR. The sequential analysis of anti-platelets (anti-GpIIbIIIa) antibodies producing B cells will be performed by means of flow cytometry and ELISPOT analysis. T cells subsets will be harvested in presence of GpIIbIIIa immunodominant peptides and and cytokines expression will be measured on supernatants on days 2 and 11 in vitro by using Luminex technology in order to characterize and distinguish TH1, TH2, TH17, TFH and Tregs subsets.

The primary outcome will be the overall response rate 1 year after inclusion defined by a platelet count > 30 x 109/L with at least a two-fold increase of the initial (pre-treatment) count. For the patients treated with rituximab as a standard of care, based on the overall expected response-rate (40-50%) and based on preliminary data on FcgammaRIIIA V/F158 distribution, the inclusion of 85 patients should be sufficient to show an association of the V158 allele and the response (b risk 20% and a 5%). Responders and non responders will be compared by non parametrical tests, a multivariate analysis will be than performed using a logistic regression model. The immunological data B and T cells subsets) obtained in both the responders and the non responders will be compared over time (To, M3, M6 and M12) by non parametrical matched tests.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Primary ITP as defined by the internation consensus on terminology (Rodeghiero et al. Blood 2009) regardless the phase of the disease (newly-diagnosed, persistent of chronic ITP)
* active ITP defined by a platelet count < 50 x 109/L at time of inclusion with indication for treatment
* Informed consent

Exclusion Criteria:

* Secondary ITP

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2012-09-28 (Actual); Primary Completion 2015-10-02 (Actual); Study Completion 2015-10-02 (Actual)

PRIMARY OUTCOMES:
The overall response rate to rituximab defined by a platelet count > 30 x 109/L with at least a two-fold increase of the initial (pre-treatment) count | 1 year after inclusion

SECONDARY OUTCOMES:
Rate of complete response (platelet count > 100 x 109/L) | at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: MICHEL Marc, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Henri Mondor Hospital, Créteil, France